CLINICAL TRIAL: NCT01371058
Title: Study of Policosanol to Improve High on Clopidogrel Platelet Reactivity After Percutaneous Coronary Stent Implantation(Spirit)
Brief Title: Study of Policosanol to Improve Platelet Reactivity After Percutaneous Coronary Stent Implantation (PCI)
Acronym: spirit
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shenyang Northern Hospital (Other)
Responsible Party: Principal Investigator, Han Yaling, Dr, Shenyang Northern Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NH-20110530
Record Dates: First submitted 2011-05-31; First posted 2011-06-10 (Estimated); Last update posted 2015-12-16 (Estimated); Status verified 2015-12

CONDITIONS: Coronary Artery Disease
Keywords: high on-treatment platelet reactivity; percutaneous coronary intervention; stent thrombosis
MeSH Terms: conditions — Coronary Artery Disease | interventions — policosanol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- routine dual antiplatelet (Active Comparator): asprin 300mg/d for 1 month followed by 100mg/d chronically； clopidogrel 75mg/d for 1year.
  Interventions: Drug: routine dual antiplatelet
- high maintenance clopidogrel (Experimental): aspirin 300mg/d for 1 month followed by 100mg/d chronically; clopidogrel 150mg/d for 1 month followed by 75mg/d for at least 1 year.
  Interventions: Drug: high maintenance clopidogrel
- policosanol plus dual antiplatelet (Experimental): asprin 300mg/d for 1 month followed by 100mg/d chronically; clopidogrel 75mg/d for at least 1 year; Policosanol 40mg/d for 6months.
  Interventions: Drug: policosanol plus dual antiplatelet

INTERVENTIONS:
Drug: high maintenance clopidogrel — clopidogrel 150 mg/d for 30 days followed by 75 mg/d for at least 1 year； aspirin 300mg/d for 1 month followed by 100mg/d chronically；
  Arms: high maintenance clopidogrel
Drug: routine dual antiplatelet — clopidogel 75mg/d for at least 1 year； aspirin 300mg/d for 1 month followed by 100mg/d chronically；
  Arms: routine dual antiplatelet
Drug: policosanol plus dual antiplatelet — aspirin 300 mg/d for 1 month followed by 100 mg/d chronically； clopidogrel 75 mg/d for at least 1 year policosanol 40mg/d for 6 months
  Arms: policosanol plus dual antiplatelet

SUMMARY:
Thrombotic event is one of the most serious complications of coronary artery disease, which often result in myocardial infarction and even death. Even according to the standard guidelines for antiplatelet therapy, there are still 6% to 15% of patients occur thrombotic events, in high-risk patients, the proportion is higher, this phenomenon is called anti-platelet drug resistance in clinical practice

The aim of this multicenter prospective, randomized, controlled study is to observed policosanol on aspirin or clopidogrel resistance in patients with platelet aggregation after Percutaneous Coronary Stent Implantation (PCI) and occurrence of platelet aggregation and short-term prognosis to find new ways to the prevention of platelet aggregation .

DETAILED DESCRIPTION:
Thrombotic event is one of the most serious complications in coronary artery disease, which often result in myocardial infarction and even death. Even according to the standard guidelines for antiplatelet therapy, there are still 6% to 15% of patients occur thrombotic events, in high-risk patients, the proportion is higher, this phenomenon is called anti-platelet drug resistance in clinical practice

ELIGIBILITY:
Inclusion Criteria:

* Patients with coronary heart disease and had received coronary stenting
* high on-treatment platelet reactivity defined as an ADP-induced platelet aggregation (by LTA)> 65% at 24 hr after clopidogrel loading (300 ~ 600mg)or 5 days after maintenance dose treatment (75mg / d)
* Informed Consent

Exclusion Criteria:

* receiving GP IIb / IIIa receptor antagonist treatment within 24h before enrollment
* using cilostazol within 7d before enrollment
* aspirin, clopidogrel or policosanol allergies
* NYHA grade III ~ IV
* planned elective coronary revascularization for multivessel coronary artery disease
* long term warfarin treatment after persistent atrial fibrillation, valve surgery or other circumstance
* Severe liver or kidney dysfunction
* Active ulcer or a history of recent gastrointestinal bleeding
* History of coagulation disorder, or recent history of active bleeding
* history of intracranial hemorrhage within 6 months
* Pregnancy
* LDL less than 70mg/dL
* Severe systemic diseases with life expectancy less than 1 year
* planned surgery within next 6 months

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Actual)
Dates: Start 2011-03; Primary Completion 2012-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
reversion rate of HPR | 30 days
  reversion was defined as platelet aggregation <65%

SECONDARY OUTCOMES:
major adverse cardiovascular events | 1 year
  including cardiac death, non-fatal myocardial infarction and target vessel revascularization
Stent thrombosis and TIMI bleeding events | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Yaling Han, MD, Principal Investigator — Shenyang Northern Hospital
Locations (1):
- The First Hospital of China Medical University, Shenyang, Liaoning, China